CLINICAL TRIAL: NCT01588197
Title: Real-Time fMRI Feedback Effects on Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR # 20270
Record Dates: First submitted 2012-02-10; First posted 2012-04-30 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Pain Control
Keywords: Pain; fMRI; real time
MeSH Terms: conditions — Pain

ARMS (2):
- ACC Real Time fMRI Feedback (Experimental): Each participant will undergo thermal pain threshold assessments ten times using the Medoc Pathway System with MRI-compatible ATS Thermode (30mmX30mm; Medoc Inc, Israel). Participants will be instructed to "focus on the thermal stimuli" for the first 5 trials, and to engage in three cognitive pain inhibition strategies (Attention/Distraction Strategy, Stimulus Quality/Severity Strategy, and the Control Strategy.
  The participants will be randomly assigned to receive Real Time fMRI Feedback of inverse activation in the rACC after each pain/rest block during the last 3 fMRI scans in the form of two simple thermometer images on the in-scanner computer display.
  Interventions: Behavioral: Attention/Distraction Strategy; Behavioral: Stimulus Quality/Severity Strategy; Behavioral: Control Strategy
- PFC Real Time fMRI Feedback (Experimental): Each participant will undergo thermal pain threshold assessments ten times using the Medoc Pathway System with MRI-compatible ATS Thermode (30mmX30mm; Medoc Inc, Israel). Participants will be instructed to "focus on the thermal stimuli" for the first 5 trials, and to engage in three cognitive pain inhibition strategies (Attention/Distraction Strategy, Stimulus Quality/Severity Strategy, and the Control Strategy. The participants will be randomly assigned to receive Real Time fMRI Feedback of inverse activation in the PFC after each pain/rest block during the last 3 fMRI scans in the form of two simple thermometer images on the in-scanner computer display.
  Interventions: Behavioral: Attention/Distraction Strategy; Behavioral: Stimulus Quality/Severity Strategy; Behavioral: Control Strategy

INTERVENTIONS:
Behavioral: Attention/Distraction Strategy — One of three Cognitive Pain Inhibition Strategies. The Participant will be instructed to attend away from the thermal stimulus (for example, to the other side of the body). Vividly imagine they are somewhere else, or engage in a high-demanding mental task such as counting backward by 7's or completing math problems to distract from the experience
Behavioral: Stimulus Quality/Severity Strategy — One of three Cognitive Pain Inhibition Strategies. The Participant will be instructed to attempt to perceive the stimulus as a neutral sensory experience rather than pain. Attempt to perceive the stimulus as low intensity rather than high intensity.
Behavioral: Control Strategy — One of three Cognitive Pain Inhibition Strategies. The Participant will be instructed to attempt to take control of their perception of the painful experience.

SUMMARY:
The purpose of this study is to determine whether real-time functional magnetic resonance imaging may be a viable treatment for chronic pain in the future.

DETAILED DESCRIPTION:
Twenty-four healthy volunteers will undergo a series of four fMRI scanning sessions wherein thermal pain stimuli will be used to elicit activation of the pain neuro-matrix. All participants will undergo thermal pain threshold testing before and after fMRI scan. Participants will also rate the painfulness and unpleasantness of the thermal stimuli applied before fMRI and after fMRI. All participants will be given prompts to apply a set of cognitive pain-control strategies. Half of the participants will receive real-time fMRI feedback of activity in the Right Anterior Cingulate Cortex (rACC) and the other half will receive real-time fMRI feedback of activity in the Prefrontal Cortex (PFC). It is hypothesized that those receiving real-time feedback of brain activity thought to be involved with analgesic effects will demonstrate greater analgesia associated with the application of the cognitive control techniques after fMRI paradigm (decreased pain intensity and unpleasantness ratings and increased thermal pain thresholds) than those who are not given feedback before fMRI paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 18-65

Exclusion Criteria:

* Clinical depression
* Anxiety
* Substance dependence or chronic pain
* Ferrous metal implants
* Cardiac pacemakers or other implanted medical devices that might be adversely impacted by the MRI scanner magnetic field

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery J Borckardt, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACC Real Time fMRI Feedback | PFC Real Time fMRI Feedback
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — No MRI | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants did not complete MRI scanning and so were not included in analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | ACC Real Time fMRI Feedback | PFC Real Time fMRI Feedback | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.65) | 24.78 (3.90) | 26.39 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 8 | 9 | 17
  Black or African American | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Average Unpleasantness
Description: All participants will undergo thermal pain threshold testing directly before (Baseline) and after MRI. Participants will be asked to rate pain unpleasantness, on a scale of 0-10, before the fMRI Paradigm (Baseline) and directly after the fMRI paradigm (after MRI).
  0="no unpleasantness" and 10="worst unpleasantness imaginable"
Time Frame: Before and After fMRI Paradigm, an average of 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACC Real Time fMRI Feedback | PFC Real Time fMRI Feedback
Number analyzed (Participants) | 9 | 9
units on a scale
  Before fMRI Paradigm | 3.75 (2.48) | 3.56 (2.22)
  After fMRI Paradigm | 3.30 (2.39) | 4.28 (2.82)

2. Primary Outcome: Average Pain Rating
Description: All participants will undergo thermal pain threshold testing directly before (Baseline) and after MRI scan.Participants will be asked to rate painfulness of the thermal stimuli applied, on a scale of 0-10, before the fMRI Paradigm (Baseline) and directly after the fMRI paradigm (after MRI). 0="no pain" and 10="worst pain imaginable"
Time Frame: Before and After fMRI Paradigm, an average of 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACC Real Time fMRI Feedback | PFC Real Time fMRI Feedback
Number analyzed (Participants) | 9 | 9
units on a scale
  Before fMRI Paradigm | 3.79 (2.20) | 3.64 (2.30)
  After fMRI Paradigm | 3.88 (2.21) | 4.43 (2.23)

3. Primary Outcome: Ability to Distract
Description: All participants will undergo thermal pain threshold testing before and after fMRI paradigm. Participants will rate the ability to distract themselves from the thermal stimuli, on a scale of 0-10, before fMRI paradigm (Baseline) and after fMRI paradigm, 0="not able to distract at all" and 10="completely able to distract". A Higher rating represents greater ability to distract from thermal pain stimuli.
Time Frame: Before and After fMRI Paradigm, an average of 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACC Real Time fMRI Feedback | PFC Real Time fMRI Feedback
Number analyzed (Participants) | 9 | 9
units on a scale
  Before fMRI Paradigm | 4.92 (1.96) | 3.83 (1.25)
  After fMRI Paradigm | 4.41 (2.15) | 4.02 (1.72)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Real Time fMRI Feedback: Each participant will undergo thermal pain threshold assessments ten times using the Medoc Pathway System with MRI-compatible ATS Thermode. They will be instructed to "focus on the thermal stimuli" for the first 5 trials, and to engage in three cognitive pain inhibition strategies (Attention/Distraction Strategy, Stimulus Quality/Severity Strategy, and the Control Strategy. Half of the participants will be randomly assigned to receive Real Time fMRI Feedback of inverse activation in the rACC and PFC after each pain/rest block.
- No Feedback: Each participant will undergo thermal pain threshold assessments ten times using the Medoc Pathway System with MRI-compatible ATS Thermode. They will be instructed to "focus on the thermal stimuli" for the first 5 trials, and to engage in three cognitive pain inhibition strategies (Attention/Distraction Strategy, Stimulus Quality/Severity Strategy, and the Control Strategy. Randomly assigned to receive no feedback in the form of two empty thermometer images on the in-scanner computer display.
Arm/Group | Real Time fMRI Feedback | No Feedback
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No